CLINICAL TRIAL: NCT03396341
Title: Responses to Genetic Risk Modifier Testing Among Women With BRCA1/2 Mutations
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Phenogen Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17-489; NCT04943250 (obsolete NCT alias)
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Genetic Testing; BRCA1/2
Keywords: BRCA1/2 Mutations; 17-489
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients receiving a positive BRCA1/2 mutation result: All interested participants will provide a saliva sample for genetic risk modifier testing, and will complete Assessment #1 questionnaires. Participants will be contacted 1 week later (+/- 1 week) to complete Assessment #2 questionnaires. Participants will be contacted 6 months (+/- 3 weeks) following the receipt of their genetic risk modifier results to complete Assessment #3 questionnaires. Participants will be encouraged to complete Assessments #2 and #3 via email using the secure, approved REDCap system
  Interventions: Other: Salvia sample; Behavioral: Questionnaires

INTERVENTIONS:
Other: Salvia sample — salvia sample
Behavioral: Questionnaires — Participants will complete Assessment #1 questionnaires. Participants will be contacted 1 week later (+/- 1 week) to complete Assessment #2 questionnaires. Participants will be contacted 6 months (+/- 3 weeks) following the receipt of their genetic risk modifier results to complete Assessment #3 questionnaires. Participants will be encouraged to complete Assessments #2 and #3 via email using the secure, approved REDCap system

SUMMARY:
The purpose of this study is to describe how women with BRCA1/2 mutations react to genetic risk modifier testing, and to examine how they make decisions about their healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Female patient, age 25 years or older (given that women under this age are not generally recommended to receive BRCA1/2 genetic testing)
* Completed full sequence or targeted genetic testing with a clinically confirmed BRCA1 or BRCA2 deleterious mutation identified
* No personal history of breast cancer
* English-fluent; the surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the surveys.

Exclusion Criteria:

* Previous receipt of any prophylactic mastectomy.
* Major psychiatric illness or cognitive impairment that in the judgment of the study investigators or study staff would preclude study participation.
* Any patients who are unable to comply with the study procedures as determined by the study investigators or study staff.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — BRACA 1/2 mutation carriers
Study Population: Potential participants (i.e., patients receiving a positive BRCA1/2 mutation result) will be identified and approached by their primary genetic counselor.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
number of patients that opt for preventive mastectomy or to pursue surveillance | 3 years
  Hierarchical level modeling (HLM) will be implemented to assess the effect of genetic risk modifier testing on Decisional Conflict Scale score (DCS), allowing for baseline effects via a random intercept.

CONTACTS AND LOCATIONS:
Overall Officials: Jada Hamilton, PhD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Dana Farber Cancer Institute (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Abramson Cancer Center at University of Pennsylvania Medical Center (Data Collection Only), Philadelphia, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm